CLINICAL TRIAL: NCT01306331
Title: A Multicenter, Open-Label, Randomized Study of the Contraceptive Efficacy and Safety of Phexxi™ (Previously Known as Amphora) Gel Compared to Conceptrol Vaginal Gel
Brief Title: Study of Contraceptive Efficacy & Safety of Phexxi™ (Previously Known as Amphora) Gel Compared to Conceptrol Vaginal Gel
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Evofem Inc. (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AMP001
Record Dates: First submitted 2011-02-28; First posted 2011-03-01 (Estimated); Results first posted 2020-07-30 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-06

CONDITIONS: Contraception
MeSH Terms: interventions — Nonoxynol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conceptrol (Active Comparator): 100 mg (4% concentration) of nonoxynol-9 in 2.5 mL volume of gel
  Interventions: Drug: Conceptrol
- Amphora (Experimental): Citric acid USP, potassium bitartrate USP, and L-lactic acid USP
  Interventions: Drug: Amphora

INTERVENTIONS:
Drug: Conceptrol — • Conceptrol® Vaginal Gel, which contains 100 mg (4% concentration) of nonoxynol-9 (N-9) in 2.5 mL volume of gel.
  Arms: Conceptrol
Drug: Amphora — • Amphora™ gel, which will be delivered in 5 mL doses, is a clear, water-based, petroleum-free gel.
  Arms: Amphora

SUMMARY:
This is a research study of a new experimental vaginal gel that helps in vaginal pH regulation and results in immobilization of spermatozoa by maintaining the normally low vaginal pH, even in the presence of semen. This vaginal gel is called Phexxi™ (previously known as Amphora) and was compared to a commercially available spermicide called Conceptrol®, which contains nonoxynol 9; commonly abbreviated as N-9. Conceptrol® can help prevent pregnancy. This study objective was to determine if this product prevents pregnancy when inserted into the vagina before intercourse.

DETAILED DESCRIPTION:
Clinical Trial Design

This is a multicenter, open-label, randomized, controlled, Phase III study of repeated use of Amphora™ gel compared to Conceptrol® Vaginal Gel as the method of contraception over seven cycles of use. In addition, there is an opportunity for Amphora™ gel subjects to continue with study treatment for up to 13 cycles of treatment upon completion of the first seven cycles of treatment.

A subset of subjects (Amphora™ gel and Conceptrol® Vaginal Gel) will undergo colposcopy at the Admission Visit and at the visits after Cycles 1, 3, and 7 (Treatment Exit). Subjects participating for 13 cycles will also undergo colposcopy after Cycles 10 and 13. Colposcopic photographs will be taken at all visits independent of presence of any suspicious areas. Any suspicious areas and clinical findings will be recorded on the colposcopy case report form. The colposcopy evaluator for the subset will be blinded regarding the treatment group of the subject. If at any time during the study the investigator deems colposcopy necessary, colposcopy will be performed on any subject and will not be limited to subjects in the colposcopy subset.

A subset of subjects (Amphora™ gel and Conceptrol® Vaginal Gel) will also have semi-quantitative cultures for E. coli and clinical yeast performed at the Admission Visit and after Cycles 1, 3, and 7 (Treatment Exit) Visits. Subjects participating for 13 cycles will also undergo the assessments after Cycles 10 and 13. Another subgroup will have quantitative vaginal cultures performed after Cycles 1 and 7 (Treatment Exit) Visits, and also after Cycle 13 for subjects participating in the extension.

Selected research centers will also recruit subjects into the subset of women 36-45 years of age at enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Be healthy women, who are sexually active, at risk for pregnancy, and desiring contraception.
* Be within the age range of 18 through 35 (inclusive) at enrollment if not in the subset of women with an age of 36-45 at enrollment (age subset at select sites).
* Be at low-risk for both human immunodeficiency virus (HIV) and sexually transmitted disease (STD) infection and currently have a single sex partner (≥ 4 months) who is also at low-risk for both HIV and STD infection.
* Have a negative urine pregnancy test prior to enrollment.
* Have normal cyclic menses with a usual length of 21 to 40 days over the last two cycles or at least one spontaneous, normal menstrual cycle (two menses) since delivery, abortion, or after discontinuing hormonal contraception/hormonal therapy.
* Be willing to accept a risk of pregnancy.
* Be willing to engage in at least two acts of heterosexual vaginal intercourse per cycle.
* Be willing to be randomized to either study treatment.
* Be willing to use the study product as the only method of contraception over the course of the study (with the exception of emergency contraception (EC)), when indicated).
* Be capable of using the study product properly and agree to observe all study directions and requirements.
* Be willing to keep a daily diary to record coital information, product use information, information about the use of other vaginal products, and sign and symptom data for both the subject and her partner.
* Agree not to participate in any other clinical trials during the course of the study with the exception of enrolling in the Amphora™ gel extension study.
* Be willing to give written informed consent to participate in the trial.

Exclusion Criteria:

* Have a history of allergy or sensitivity to spermicides or products containing N-9 (nonoxynol-9).
* Have had three or more urinary tract infections (UTIs) in the past year.
* Have a UTI by urine culture, symptomatic yeast vaginitis, or symptomatic bacterial vaginosis diagnosed by wet mount unless treated and proof of cure is documented.
* Have a history of any recurrent vaginal infections/disorders (either less than or equal to four times in the past year or less than or equal to three times in the previous six months).
* Be pregnant, have a suspected pregnancy, or desire to become pregnant during the course of the study.
* Have a history of infertility or of conditions that may lead to infertility, without subsequent intrauterine pregnancy.
* Have any contraindications to pregnancy (medical condition) or chronic use of medications for which significant evidence of fetal risk exists.
* Have had more than one sexual partner in the last four months.
* Have shared injection drug needles in the past unless has a negative HIV test at least six weeks since last use.
* Have or have been suspected to have HIV infection.
* Have been diagnosed with genital herpes simplex virus (HSV), with the first occurrence (initial episode) within three months prior to screening.
* Have three or more outbreaks of HSV within the last year.
* Have evidence of Chlamydia trachomatis or Neisseria gonorrhoeae unless she and her partner complete treatment and proof of cure is documented.
* Have been diagnosed with any other STDs in the six months prior to the Randomization Visit (with the exception of human papillomavirus (HPV), trichomonas, gonorrhea, adn Chlamydia).
* Be lactating or breastfeeding.
* Have any clinically significant abnormal vaginal bleeding or spotting within the month prior to screening.
* Have any clinically significant abnormal finding on pelvic examination or baseline labs, which in the view of the investigator, precludes her from participating in the trial.
* Have clinically significant signs of vaginal or cervical irritation on pelvic examination.
* Have had vaginal or cervical biopsy or vaginal surgery within three months prior to screening (with the exception of cervical biopsies performed for eligibility determination).
* Have used vaginal or systemic antibiotics or antifungals within 14 days prior to screening or enrollment/randomization, with the exception of systemic antibiotics taken for a UTI and trichomonas diagnosed at screening. Subjects should not have used systemic antibiotics prescribed at the Screening Visit for a UTI within seven days of the enrollment/randomization visit.
* Have had a Depo-Provera® injection in the ten months prior to enrollment.
* Have an abnormal Pap test based on the following criteria:
* Pap test in the past 15 months with ASC-US unless:
* less than 21 years of age;
* a repeat Pap test at least six months later was normal;
* reflex HPV testing was performed and was negative for high-risk HPV; or
* a colposcopy (with or without biopsy) found no evidence of dysplasia requiring treatment or treatment was performed and follow-up at least six months after the treatment showed no evidence of disease;
* Pap test in the past 15 months with LSIL unless:
* less than 21 years of age;
* a colposcopy (with or without biopsy) found no evidence of dysplasia requiring treatment or treatment was performed and follow-up at least six months after the treatment showed no evidence of disease;
* Pap test in the past 15 months with ASC-H, atypical glandular cells, or HSIL unless colposcopy and/or treatment was performed and follow-up at least six months after the colposcopy and/or treatment showed no evidence of disease;
* Pap test in the past 15 months with malignant cells.
* Consume (on average) greater than three drinks of an alcoholic beverage per day.
* Have a past history (within 12 months) or current history which, in the PI's judgment, constitutes of drug abuse (recreational, prescription, or over-the-counter (OTC)).
* Have taken an investigational drug or used an investigational device within the past 30 days.
* Have issues or concerns (in the judgment of the investigator) that may compromise the safety of the subject or confound the reliability of compliance and information acquired in this study.

In addition, in order to be eligible to participate in the trial, potential subjects must state that, to her best knowledge, her sexual partner meets the following criteria:

* Is not infertile.
* Has had untreated chlamydia or gonorrhea in the past six months.
* Has not had more than one sexual partner in the past four months.
* Has no history of allergy or sensitivity to spermicides or products containing N-9.
* Has not been previously diagnosed with or suspected of HIV infection unless he has subsequently had a negative HIV test.
* Has not been known to have engaged in homosexual intercourse in the past five years unless he has had negative HIV test results since then.
* Has not shared injection drug needles in the past unless he has had a negative HIV test at least six weeks since last use.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3389 (Actual)
Dates: Start 2011-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Culwell, MD, Study Director — Evofem Inc.
Locations (52):
- United States (41):
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - Advanced Clinical Research Institute, Anaheim, California
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - California Family Health Council, Inc., Berkeley, California
  - California Family and Health Council, Inc., LA, Los Angeles, California
  - California Family Health Council, Los Angeles, California
  - Women's Health Care, San Diego, California
  - Downtown Women's Healthcare, Denver, Colorado
  - Planned Parenthood of the Rocky Mountains, Denver, Colorado
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Meridien Research, Bradenton, Florida
  - Avail Clinical Reseach, DeLand, Florida
  - Altus Research, Lake Worth, Florida
  - Miami Research Associates, Miami, Florida
  - Segal Institute for Clinical Research, North Miami, Florida
  - Meridien Research, St. Petersburg, Florida
  - Comprehensive Clinical Trials, West Palm Beach, Florida
  - Soapstone Center for Clinical Research, Decatur, Georgia
  - Rosemark WomenCare Specialist, Idaho Falls, Idaho
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Johns Hopkins Community Physicians, Baltimore, Maryland
  - Impact Clinical Trials, Las Vegas, Nevada
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - NYU Medical Center Family Planning, New York, New York
  - Columbia University Medical Center, Division of Family Planning, New York, New York
  - Eastern Carolina Women's Center, New Bern, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Planned Parenthood of Northeast Ohio, Cleveland, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - University of Pennsylvania Medical Center, Reproductive Research Unit, Philadelphia, Pennsylvania
  - Philadelphia Clinical Research, Philadelphia, Pennsylvania
  - Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - Advanced Research Associates, Corpus Christi, Texas
  - Practice Research Organization, Dallas, Texas
  - UT Southwestern Medical Center - Dept. of OB/GYN, Dallas, Texas
  - TMC Life Research, Inc, Houston, Texas
  - MacArthur OB/GYN, Irving, Texas
  - Jean Brown Research, Salt Lake City, Utah
  - Women's Clinical Research Center, Seattle, Washington
- Russia (11):
  - Kazan State Medical University, Kazan', Republic Tatarstan
  - State Budgetary Institution fo Rostov region "Parinatal Center", Rostov-on-Don, Rostov Oblast
  - Moscow Regional Research Institute of Obstetrics and Gynecology, Moscow
  - City Clinical Hospital #13, Moscow
  - City Clinical Hospital #31, Moscow
  - First Moscow State Medical University named after IM Sechenov, Moscow
  - Maternity Hospital #17, Saint Petersburg
  - Medical Center "Prime-Rose"LLC, Saint Petersburg
  - The DO Ott Research Institute of Obstetrics and Gynecology, Saint Petersburg
  - Hospital OrCli, Saint Petersburg
  - Ural Scientific Research Institution of Maternity and Child Protection, Yekaterinburg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy, sexually active women at risk of pregnancy who desired contraception, aged 18 to 35 years, with a single male sex partner, of which both partners were at low risk for HIV and sexually transmitted disease (STD) infection. Subjects were required to have regular, normal, cyclic menses with a usual length of 21 to 40 days.
Pre-assignment Details: The study had 65 randomized screen failures and were not included in the ITT population due to being accidentally randomized (30 randomized to Amphora™ Gel and 35 to Conceptrol®).
Period: Overall Study
Arm/Group | Conceptrol | Amphora
Started | 1659 | 1665
Completed | 758 | 788
Not Completed | 901 | 877
Not completed — Adverse Event | 28 | 25
Not completed — Lost to Follow-up | 321 | 323
Not completed — Physician Decision | 26 | 22
Not completed — Pregnancy | 136 | 151
Not completed — Protocol Violation | 154 | 124
Not completed — Withdrawal by Subject | 163 | 152
Not completed — Not sexually active | 29 | 28
Not completed — Meth. no longer prim. meth. birth cntrl | 10 | 20
Not completed — Other | 34 | 32

BASELINE CHARACTERISTICS:
Population: Intent-Treat-Population - subjects randomized into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Conceptrol | Amphora | Total
Number analyzed (Participants) | 1659 | 1665 | 3324
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.6 (5.7) | 27.6 (5.6) | 27.6 (5.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1659 | 1665 | 3324
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 385 | 392 | 777
  Not Hispanic or Latino | 1274 | 1272 | 2546
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 14 | 23
  Asian | 45 | 36 | 81
  Native Hawaiian or Other Pacific Islander | 13 | 9 | 22
  Black or African American | 464 | 471 | 935
  White | 1030 | 1031 | 2061
  More than one race | 98 | 102 | 200
  Unknown or Not Reported | 0 | 2 | 2
BMI Category at Enrollment (kg/m2) [Count of Participants; unit: Participants]
  Underweight (<18.5) | 75 | 83 | 158
  Normal (18.5 - 24.9) | 672 | 640 | 1312
  Overweight (25.0 - 29.9) | 369 | 392 | 761
  Obese (>30.0) | 539 | 548 | 1087
BMI at Enrollment (kg/m2) [Mean (Standard Deviation); unit: kg/m2] | 27.76 (7.98) | 27.91 (7.95) | 27.83 (7.97)

OUTCOME MEASURES:

1. Primary Outcome: 6-Month (183 Days) Cumulative Pregnancy Percentage
Description: The primary endpoint was the evaluation of contraceptive efficacy over six months (183 days) of Amphora™ Gel use when compared to Conceptrol® Vaginal Gel. Kaplan-Meier methods were used to estimate the six-month cumulative pregnancy percentage of women in the MITT population by treatment group
Time Frame: 183 days
Population: mITT Population - ITT subjects whose diaries indicated they had at least one episode of coitus while using the assigned study product (also referred as "Typical-Use"), between 18 to 35 years of age (inclusive) at enrollment, had at least 1 cycle without any backup contraception or EC, and for whom there was at least one report of pregnancy status.
Measure: Mean (95% Confidence Interval); unit: pregnancy percentage
Arm/Group | Conceptrol | Amphora
Number analyzed (Participants) | 1281 | 1259
pregnancy percentage | 10.0 [8.1 to 11.9] | 10.5 [8.6 to 12.3]
Statistical Analysis 1: Comparison: Conceptrol vs Amphora; The primary hypothesis test was performed using 95% confidence interval for the difference in cumulative pregnancy rates between the treatment arms. If the upper bound for the confidence interval of the difference was < 5.5, then the null hypothesis would be rejected; Test type: Non-Inferiority — If the upper bound for the confidence interval of the difference was < 5.5, then the null hypothesis would be rejected; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-2.2 to 3.2]

2. Secondary Outcome: 6-Month (183 Days) Cumulative Pregnancy Percentage for Subjects With Perfect Use
Description: Perfect use contraceptive efficacy over six months (183 days) of Amphora™ Gel use when compared to Conceptrol® Vaginal Gel. Kaplan-Meier methods were used to estimate the six-month cumulative pregnancy percentage of women in the efficacy evaluable (EE) population by treatment group
Time Frame: 183 days
Population: EE populations - a subset of the MITT population that includes only subjects with at least one EE cycle, where an EE cycle is a cycle where the diaries indicated they used the product correctly for every act of intercourse in the cycle.
Measure: Mean (95% Confidence Interval); unit: pregnancy percentage
Arm/Group | Conceptrol | Amphora
Number analyzed (Participants) | 1161 | 1161
pregnancy percentage | 4.2 [2.8 to 5.6] | 4.1 [2.7 to 5.4]

ADVERSE EVENTS:
Time Frame: 183 days
Description: Any untoward medical occurrence in a subject that has been treated with study drug; the untoward medical occurrence did not necessarily have to have a causal relationship with the study treatment; In reference to the total number of participants at risk in the adverse events module, the # at risk was limited to the # of ITT subjects who used at least 1 dose of drug.
Arm/Group | Conceptrol | Amphora
All-Cause Mortality (participants affected / at risk) | 0/1477 | 0/1458
Serious Adverse Events (participants affected / at risk) | 19/1477 | 11/1458
Other Adverse Events (participants affected / at risk) | 857/1477 | 793/1458
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Conceptrol (N=1477) | Amphora (N=1458)
Wolff-Parkison-White syndrome (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Non-cardiac chest pain (Gastrointestinal disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 1
Appendicitis (Infections and infestations) | 1 | 0
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Kidney Infection (Infections and infestations) | 1 | 0
Post procedural sepsis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 2 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 2
Investigation (Investigations) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Migraine (Nervous system disorders) | 0 | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 3 | 1
Ovarian rupture (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Gastrectomy (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Conceptrol (N=1477) | Amphora (N=1458)
Urinary Tract Infection (Infections and infestations) | 193 | 140
Vaginitis Bacterial (Infections and infestations) | 170 | 160
Vulvovaginal Mycotic (Infections and infestations) | 168 | 156
Headache (Nervous system disorders) | 80 | 96
Vulvovaginal Pruritus (Reproductive system and breast disorders) | 76 | 55
Nasopharyngitis (Infections and infestations) | 48 | 76
Vulvovaginal Discomfort (Reproductive system and breast disorders) | 53 | 42
Vulvovaginal (Infections and infestations) | 46 | 45
Vulvovaginal Burning Sensation (Reproductive system and breast disorders) | 41 | 49
Vaginal Discharge (Reproductive system and breast disorders) | 46 | 43
Dysmenorrhoea (Reproductive system and breast disorders) | 34 | 33
nfluenza (Infections and infestations) | 20 | 37
Smear Cervix Abnormal (Investigations) | 29 | 21
Dysuria (Renal and urinary disorders) | 30 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes